CLINICAL TRIAL: NCT01469286
Title: Transcutaneous Electroacupuncture for Gastroparesis
Acronym: TEA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Transtimulation Research, Inc (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); University of Mississippi Medical Center (Other); Texas Tech University Health Sciences Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: TEA-Gastroparesis; R43AT004489 (NIH)
Record Dates: First submitted 2011-11-08; First posted 2011-11-10 (Estimated); Last update posted 2017-05-01 (Actual); Status verified 2017-04

CONDITIONS: Diabetic Gastroparesis
Keywords: delayed gastric emptying; nausea; vomiting; abdominal discomfort
MeSH Terms: conditions — Gastroparesis; Nausea; Vomiting

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TEA (Active Comparator): Needleless electroacupuncture at ST36 and PC6
  Interventions: Device: TEA
- Sham-TEA (Placebo Comparator): Needleless acupuncture at sham-points
  Interventions: Device: Sham-TEA

INTERVENTIONS:
Device: TEA — Electroacupuncture at ST36
  Arms: TEA
Device: Sham-TEA — Electroacupuncture at sham-points
  Arms: Sham-TEA

SUMMARY:
Gastroparesis is a common disease defined as delayed emptying of the stomach. It is present in at least 20% of about 150 million patients with diabetes worldwide and in more than 20% of patients with functional dyspepsia that affects about 10%-25% of the general population. Gastroparesis is a refractory disease with a lack of therapeutic options. Common symptoms of gastroparesis include nausea, vomiting, early satiety and abdominal bloating.

Electroacupuncture (EA) is a combined procedure with acupuncture and electrical current stimulation instead of manual manipulations of the needles. Recent studies in our lab with EA or transcutaneous EA (TEA) have suggested a therapeutic role of EA or TEA for gastric motility disorders. Improvement has been observed with EA or TEA in gastric emptying as well as dyspeptic symptoms. In this project, a micro-stimulator is designed and developed for the TEA therapy. The micro-stimulator is small enough so that it can be attached to the skin next to the stimulation electrodes and therefore the patient can resume normal daily activity while being treated by TEA. This is not only attractive but also more effective since TEA can be performed more often and for longer durations.

This exploratory project is designed to study the feasibility, efficacy and certain mechanisms of the proposed method of "wireless" TEA in patients with gastroparesis. Firstly the feasibility of the chronic use the proposed micro-stimulator will be studied. Secondly, the efficacy of the TEA in improving delayed gastric emptying and symptoms of gastroparesis will be investigated in a double-blinded crossover design in patients with diabetic or idiopathic gastroparesis. Thirdly, possible mechanisms involving pathogeneses of gastroparesis with TEA will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* At least one severe gastroparetic symptom or two moderate gastroparetic symptoms (see assessment of gastroparetic symptoms);
* Abnormal gastric emptying defined as more than 10% of gastric retention at 4 hrs after a standard solid meal (see below) during the past 3 months;
* Males and females between ages 18-65 yrs;
* Subjects with high probability for compliance and completion of the study.
* Upper endoscopy or upper GI within last 2 years showing no evidence of gastric bezoar, stricture, or peptic ulcer.
* Diabetes.

Exclusion Criteria:

1) History of gastric bezoar or diverticulitis. 2) Severe daily abdominal pain requiring medications for relief. 3) Severe weight loss, greater than 10 lbs over the preceding 2 months. 4) Uncontrolled diabetes with a hemoglobin A1C greater than 10. 5) Excessively delayed gastric emptying time: more than 90% of a standard meal retained after 2 hours. 6) Previous gastro-esophageal surgery including vagotomy, fundoplication, gastric bypass, ulcer surgery. 7) Prior GI surgery except for uncomplicated appendectomy and laparoscopic cholecystectomy; 8) Surgery within the past 3 months. 9) Female of childbearing age who is not practicing birth control and/or is pregnant or lactating. (Confirm with urine pregnancy test). 10) Those who have been treated with acupuncture or those who are familiar with acupuncture points. 11). Allergic to Ensure, strawberry jam and eggs.

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2010-03; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
gastroparesis symptoms | 4 weeks
  Gastroparetic symptom questionnaire will use the previously validated gastroparesis cardinal symptom index (GCSI), including 9 symptoms: nausea (feeling sick to your stomach as if you were going to vomit or throw up), retching (heaving as if to vomit, but nothing comes up), vomiting, stomach fullness, not able to finish a normal sized meal, feeling excessively full after meals, loss of appetite, bloating (feeling like you need to loose your clothes) and stomach or belly visibly larger. Each symptom will be graded from 0 to 5 (none, very mild, mild, moderate, severe and very severe).

SECONDARY OUTCOMES:
Gastric emptying | 4 weeks
  Gastric emptying of a solid meal.

CONTACTS AND LOCATIONS:
Overall Officials: Jiande Chen, PhD, Principal Investigator — Transtimulation Research, Inc
Locations (2):
- United States (2):
  - University of Mississippi, Jackson, Mississippi
  - Texas tech university health science center, El Paso, Texas